CLINICAL TRIAL: NCT06521697
Title: Anesthetic-sparing and Renal Protection Effects of Minimal-flow Sevoflurane Anesthesia and Multimodal Analgesia Using a Mixture of Dexmedetomidine-ketamine-lidocaine in Head and Neck Cancer Patients With Free Flap Microvascular Surgery
Brief Title: Effects of Minimal-Flow Sevoflurane and Multimodal Analgesia in Head and Neck Cancer Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202403100MIND
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer; Anesthesia; Renal Protection; Acute Kidney Injury; Multimodal Analgesia
Keywords: Greenhouse gas; Carbon emissions; Acute kidney injury; Multimodal analgesia; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: This study is a single-center, prospective, 2x2 factorial randomized controlled trial designed to evaluate the anesthetic-sparing and renal protection effects of minimal-flow (intervention 1) sevoflurane anesthesia combined with multimodal analgesia (intervention 2) in head and neck cancer patients undergoing free flap microvascular surgery. Participants will be randomly assigned to one of four groups:
  Fresh gas flow at 0.5 L/min with dexmedetomidine-ketamine-lidocaine mixture. Fresh gas flow at 0.5 L/min with normal saline. Fresh gas flow at 1.0 L/min with dexmedetomidine-ketamine-lidocaine mixture. Fresh gas flow at 1.0 L/min with normal saline.
  The study uses triple blinding (participant, care provider, investigator) to ensure unbiased results. The primary purpose of the study is treatment, aiming to reduce anesthetic usage and assess renal protection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a triple-blinding approach to ensure unbiased results. The participants, care providers (including anesthesiologists and nurses), and investigators are all blinded to the group assignments. Randomization envelopes containing the treatment allocation will be prepared and sealed by a research assistant who is not involved in patient care or data collection.
  At the time of surgery, the envelope will be opened by a designated anesthesia nurse who will prepare the study medication (either the dexmedetomidine-ketamine-lidocaine mixture or normal saline) according to the randomization. The medication will be labeled identically to maintain blinding and administered via continuous infusion during anesthesia. Fresh gas flow settings will be adjusted according to the randomization and indicated by a concealed flow meter display.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (HL-D) (Experimental): Fresh gas flow at 0.5 L/min with dexmedetomidine-ketamine-lidocaine mixture
  Interventions: Drug: Multimodal analgesia using dexmedetomidine-ketamine-lidocaine mixture; Device: Minimal flow sevoflurane
- Group 2 (HL-ND) (Experimental): Fresh gas flow at 0.5 L/min with placebo normal saline
  Interventions: Device: Minimal flow sevoflurane
- Group 3 (L-D) (Experimental): Fresh gas flow at 1.0 L/min with dexmedetomidine-ketamine-lidocaine mixture
  Interventions: Drug: Multimodal analgesia using dexmedetomidine-ketamine-lidocaine mixture
- Group 4 (L-ND) (No Intervention): Fresh gas flow at 1.0 L/min with placebo normal saline

INTERVENTIONS:
Drug: Multimodal analgesia using dexmedetomidine-ketamine-lidocaine mixture — Multimodal analgesia using dexmedetomidine-ketamine-lidocaine mixture vs placebo normal saline
  Other Names: Multimodal analgesia
  Arms: Group 1 (HL-D); Group 3 (L-D)
Device: Minimal flow sevoflurane — Minimal flow sevoflurane anesthesia (0.5 L/min) vs low flow sevoflurane (1 L/min)
  Arms: Group 1 (HL-D); Group 2 (HL-ND)

SUMMARY:
This study evaluates the anesthetic-sparing and renal protection effects of minimal-flow sevoflurane anesthesia combined with multimodal analgesia using dexmedetomidine, ketamine, and lidocaine in head and neck cancer patients undergoing free flap microvascular surgery. The 2x2 factorial randomized controlled trial aims to compare sevoflurane usage and renal function changes with different fresh gas flow rates and multimodal analgesia.

DETAILED DESCRIPTION:
This study investigates the anesthetic-sparing and renal protection effects of minimal-flow sevoflurane anesthesia combined with a multimodal analgesia strategy using dexmedetomidine, ketamine, and lidocaine in head and neck cancer patients undergoing free flap microvascular surgery. The trial employs a 2x2 factorial randomized controlled design to evaluate the effectiveness of different fresh gas flow rates and multimodal analgesia on sevoflurane usage and renal function.

Background and Significance:

Sevoflurane, a widely used anesthetic for prolonged surgeries, significantly contributes to healthcare-related greenhouse gas emissions. Reducing fresh gas flow during anesthesia effectively minimizes anesthetic usage, but concerns about potential renal damage hinder its clinical application. Recent studies show that sevoflurane enhances renal sympathetic nerve activity, leading to decreased renal blood flow and increased risks of acute kidney injury, particularly when coupled with factors like low blood pressure.

Multi-modal analgesia combining drugs like dexmedetomidine, ketamine, and lidocaine has emerged as a trend in anesthesiology. These drugs not only reduce sevoflurane usage but may also counteract its renal effects. This project aims to investigate the renal protective effects and anesthetic reduction potential of a multi-modal analgesia strategy in head and neck cancer surgeries.

Study Objectives:

To evaluate the anesthetic-sparing effect of minimal-flow sevoflurane anesthesia (0.5 L/min) combined with dexmedetomidine-ketamine-lidocaine multimodal analgesia.

To assess the renal protection effects of dexmedetomidine-ketamine-lidocaine multimodal analgesia during minimal-flow sevoflurane anesthesia.

To examine the safety and other potential effects (e.g., hemodynamic stability, postoperative cognitive function) of the combined anesthesia strategy.

Methods:

The study will be conducted at National Taiwan University Hospital and will involve adult patients (18-99 years) scheduled for head and neck cancer tumor resection and free flap reconstruction surgery. Patients will be randomized into four groups in a 2x2 factorial design:

Group 1 (HL + D): Fresh gas flow at 0.5 L/min with dexmedetomidine-ketamine-lidocaine mixture.

Group 2 (HL): Fresh gas flow at 0.5 L/min with normal saline. Group 3 (D): Fresh gas flow at 1.0 L/min with dexmedetomidine-ketamine-lidocaine mixture.

Group 4 (Control): Fresh gas flow at 1.0 L/min with normal saline. The dexmedetomidine-ketamine-lidocaine mixture will be continuously infused from the induction of anesthesia until the end of surgery. Fresh gas flow settings will be maintained using the EtControl function of the GE Aisys CS2 anesthesia machine. Anesthetic depth and hemodynamic parameters will be monitored throughout the procedure.

Data Collection:

Primary Outcome Measures: Sevoflurane usage (mL/h) and changes in renal function (serum renin, AVP levels, urine KIM-1, NGAL levels).

Secondary Outcome Measures: Incidence of acute kidney injury, hemodynamic stability, postoperative pain scores, length of hospital stay, and postoperative cognitive function.

Blood and urine samples will be collected at four time points: before anesthesia induction, upon arrival in the ICU, 24 hours post-surgery, and 48 hours post-surgery. Clinical data, including demographic information, surgical details, anesthetic drug usage, hemodynamic parameters, and postoperative outcomes, will also be recorded.

Statistical Analysis:

Data will be analyzed using appropriate statistical methods, including Student's t-test, Mann-Whitney U test, Chi-square test, Fisher's exact test, and multivariate analysis of variance (MANOVA). Statistical significance will be defined as p < 0.05.

Potential Challenges and Solutions:

Potential challenges include patient recruitment and adherence to protocol. To mitigate these, the study will involve experienced anesthesiologists and research staff who will ensure proper patient selection and protocol compliance.

Expected Outcomes:

The study aims to propose a feasible strategy to mitigate sevoflurane's renal effects, crucial for patients at risk of acute kidney injury. It also seeks to validate that minimal fresh gas flow (0.5 L/min) during sevoflurane anesthesia, coupled with multimodal analgesia, reduces sevoflurane usage, saving costs and contributing to carbon reduction. Additionally, the study will explore the potential protective effects of the multimodal analgesia strategy on other organs during prolonged surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99 years
* Scheduled for head and neck cancer tumor resection and free flap reconstruction surgery

Exclusion Criteria:

* Preoperative tracheostomy
* History of previous head and neck cancer tumor resection
* Anemia (hematocrit <30% or recent transfusion)
* Hypertension on ACEI/ARB medications
* Significant medical conditions (e.g., NYHA class 3 or 4 heart failure, eGFR <60 ml/min/1.73 m², Child B or C liver failure, severe respiratory disorders, pre-existing cognitive impairment)
* ASA physical status 4 or 5
* Allergies to sevoflurane, dexmedetomidine, ketamine, or lidocaine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sevoflurane usage (mL/h) | Intraoperative period
  Volatile anesthetic consumption hourly
Renal function | Perioperative period
  Changes in renal function (serum renin, AVP levels, urine KIM-1, NGAL levels)

SECONDARY OUTCOMES:
Acute kidney injury | Perioperative period
  Incidence of acute kidney injury
Hemodynamic stability_1 | Intraoperative period
  Hemodynamic stability, present as heart rate fluctuation
Hemodynamic stability_2 | Intraoperative period
  Hemodynamic stability, present as blood pressure fluctuation
Hemodynamic stability_3 | Intraoperative period
  Hemodynamic stability, present as vasoactive drug amount of usage
Postoperative analgesic effect_1 | Perioperative period
  Postoperative pain scores (VAS)
Postoperative analgesic effect_2 | Perioperative period
  Postoperative analgesic consumption
Length of hospital stay | Perioperative period
  Length of hospital stay after surgery
Cognitive function | Perioperative period
  Incidence of postoperative cognitive dysfunction using Confusion Assessment Method-Intensive Care Unit (CAM-ICU)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hui Hung, MD, Principal Investigator — National Taiwan University Hosital